CLINICAL TRIAL: NCT03469570
Title: A Validation of the Assisted Fluid Management Feature
Brief Title: Assisted Fluid Management IDE Study
Acronym: AFM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-011
Record Dates: First submitted 2018-03-12; First posted 2018-03-19 (Actual); Results first posted 2024-11-08 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2019-05

CONDITIONS: Non-Cardiac/ Non-Thoracic Surgery; Abdominal Surgery; Pelvic Surgery; Major Peripheral Vascular Surgery
Keywords: Non-Cardiac; Non-Thoracic; Fluid Management; Perioperative Goal Directed Therapy
MeSH Terms: interventions — Microscopy, Atomic Force

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Assisted Fluid Management (Experimental): Subjects enrolled in the validation study will have their fluid management decisions guided by the Acumen™ Assisted Fluid Management Feature. The Principal Investigator will accept or decline fluid recommendations.
  Interventions: Device: EV1000 Clinical Platform with Assisted Fluid Management (AFM) Feature

INTERVENTIONS:
Device: EV1000 Clinical Platform with Assisted Fluid Management (AFM) Feature — Subjects enrolled in the validation study will have their fluid management decisions guided by the AFM Feature.

SUMMARY:
The primary objective of this study is to evaluate the performance of the Acumen™ Assisted Fluid Management (AFM) Feature in its ability to predict a subject's fluid responsiveness.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the performance of the Acumen™ Assisted Fluid Management (AFM) Feature in its ability to predict a subject's fluid responsiveness.

Subjects enrolled in the validation study will have their fluid management decisions guided by the AFM Feature.

ELIGIBILITY:
Inclusion Criteria:

* Be ≥ 18 years of age
* Abdominal, pelvic, major peripheral vascular surgery expected to last >2 hours post anesthesia induction
* Participate or have authorized representative participate in the Informed Consent process and sign/date the IRB approved informed consent form.

Exclusion Criteria:

* Are < 18 years of age
* Emergent or cardiovascular surgical procedure
* Are pregnant
* Participation in any other drug, device, or biologic study concomitantly, or within the last 30 days (which may clinically interfere with this Clinical Study)
* Refusal of patient or authorized representative to sign consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Actual)
Dates: Start 2018-04-19 (Actual); Primary Completion 2018-12-21 (Actual); Study Completion 2019-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tina Abdelnour, MS, BSN, Study Director — Edwards Lifesciences
Locations (10):
- United States (10):
  - Loma Linda Health University, Loma Linda, California
  - University of California, Davis, Sacramento, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Stony Brook Medicine, Stony Brook, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Greenville Health System, Greenville Memorial Hospital, Greenville, South Carolina
  - The University of Texas Southwestern at Clements, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weiser TG, Regenbogen SE, Thompson KD, Haynes AB, Lipsitz SR, Berry WR, Gawande AA. An estimation of the global volume of surgery: a modelling strategy based on available data. Lancet. 2008 Jul 12;372(9633):139-144. doi: 10.1016/S0140-6736(08)60878-8. Epub 2008 Jun 24. PMID 18582931

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Assisted Fluid Management
Started | 330
Completed | 307
Not Completed | 23

BASELINE CHARACTERISTICS:
Population: Arterial Pressure Monitoring (enrolled) N=330. Two pilot subjects were permitted per site for training purposes N=16. Pivotal Cohort (Safety) N=314.
Arm/Group | Assisted Fluid Management
Number analyzed (Participants) | 330
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Arterial Pressure Monitoring (enrolled) N=330. Two pilot subjects were permitted per site for training purposes N=16. Pivotal Cohort (Safety) N=314.
  years
    number analyzed (Participants) | 314
    (all) | 66 [59 to 73]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Arterial Pressure Monitoring (enrolled) N=330. Two pilot subjects were permitted per site for training purposes N=16. Pivotal Cohort (Safety) N=314.
  Participants
    number analyzed (Participants) | 314
    Female | 131
    Male | 183
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Measure Analysis Population Description: Arterial Pressure Monitoring (enrolled) N=330. Two pilot subjects were permitted per site for training purposes N=16. Pivotal Cohort (Safety) N=314.
  Participants
    Rance and Ethnicity: number analyzed (Participants) | 314
    Rance and Ethnicity: Asian | 2
    Rance and Ethnicity: African American | 22
    Rance and Ethnicity: White | 284
    Rance and Ethnicity: Other | 5
    Rance and Ethnicity: Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of the Assisted Fluid Management Feature
Description: Stroke volume change meeting the clinician-selected fluid strategy
Time Frame: 30 Day follow-up
Measure: Count of Participants; unit: Participants
Arm/Group | Assisted Fluid Management
Number analyzed (Participants) | 314
Participants | 307

ADVERSE EVENTS:
Time Frame: 9 Months
Arm/Group | Assisted Fluid Management
All-Cause Mortality (participants affected / at risk) | 0/314
Serious Adverse Events (participants affected / at risk) | 88/314
Other Adverse Events (participants affected / at risk) | 226/314
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Assisted Fluid Management (N=314)
Cardiac arrest (Cardiac disorders) | 2
Arrhythmia (Cardiac disorders) | 5
Asthenia (General disorders) | 1
Complication associated with device (General disorders) | 2
Oedema (General disorders) | 1
Pain (General disorders) | 1
Pyrexia (General disorders) | 3
Biliary colic (Hepatobiliary disorders) | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Leukocytosis (Blood and lymphatic system disorders) | 1
Syncope (Cardiac disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Colites (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 1
Intestinal ischaemia (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 3
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Malaena (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Pancreatitis necrotising (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Graft infection (Infections and infestations) | 1
Ophthalmic herpes simplex (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Pancreatic abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Purulent discharge (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 8
Streptococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 3
Wound infection (Infections and infestations) | 10
Anastomotic leak (Injury, poisoning and procedural complications) | 4
Cement embolism (Injury, poisoning and procedural complications) | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 1
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 3
Procedural haemorrhage (Injury, poisoning and procedural complications) | 2
Stoma site discomfort (Injury, poisoning and procedural complications) | 1
Stoma site ischaemia (Injury, poisoning and procedural complications) | 1
Blood culture positive (Investigations) | 1
Oxygen saturation decreased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 1
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Intracranial hypotension (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Device occlusion (Product Issues) | 1
Acute kidney injury (Renal and urinary disorders) | 8
Hydronephrosis (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 1
Vesical fistula (Renal and urinary disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Abscess drainage (Surgical and medical procedures) | 1
Deep vein thrombosis (Vascular disorders) | 4
Distributive shock (Vascular disorders) | 1
Haematoma (Vascular disorders) | 4
Hypotension (Vascular disorders) | 4
Peripheral artery thrombosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Shock haemorrhagic (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Assisted Fluid Management (N=314)
Anaemia (Blood and lymphatic system disorders) | 55
Leukocytosis (Blood and lymphatic system disorders) | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Arrhythmia (Cardiac disorders) | 13
Atrial fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Sinus bradycardia (Cardiac disorders) | 1
Syncope (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 7
Diplopia (Eye disorders) | 1
Eye Swelling (Eye disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Ascites (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 4
Crohn's disease (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Duodenal ulcer (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Haematemesis (Gastrointestinal disorders) | 2
Haematochezia (Gastrointestinal disorders) | 2
Ileus paralytic (Gastrointestinal disorders) | 7
Impaired gastric emptying (Gastrointestinal disorders) | 2
Intestinal ischaemia (Gastrointestinal disorders) | 2
Intestinal obstruction (Gastrointestinal disorders) | 4
Intra-abdominal fluid collection (Gastrointestinal disorders) | 1
Jejunal perforation (Gastrointestinal disorders) | 1
Lower gastrointestinal perforation (Gastrointestinal disorders) | 1
Melaena (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 12
Obstruction gastric (Gastrointestinal disorders) | 1
Oedematous pancreatitis (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 2
Pancreatitis necrotising (Gastrointestinal disorders) | 1
Peritoneal haemorrhage (Gastrointestinal disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 13
Vomiting projectile (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Catheter site ischaemia (General disorders) | 1
Complication associated with device (General disorders) | 3
Hypothermia (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Oedema (General disorders) | 13
Pain (General disorders) | 3
Pyrexia (General disorders) | 6
Bile duct obstruction (Hepatobiliary disorders) | 1
Bile duct stenosis (Hepatobiliary disorders) | 1
Biliary colic (Hepatobiliary disorders) | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1
Abdominal infection (Infections and infestations) | 2
Abscess (Infections and infestations) | 1
Bacteraemia (Infections and infestations) | 5
Bacterial disease carrier (Infections and infestations) | 1
Bronchitis viral (Infections and infestations) | 1
Tenderness (General disorders) | 1
Cellulitis (Infections and infestations) | 2
Clostridium difficile colitis (Infections and infestations) | 1
Device related sepsis (Infections and infestations) | 1
Diverticulitis (Infections and infestations) | 1
Gangrene (Infections and infestations) | 1
Graft infection (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Ophthalmic herpes simplex (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pancreatic abscess (Infections and infestations) | 1
Peritonitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 8
Purulent discharge (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 1
Pyuria (Infections and infestations) | 1
Scrotal infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 9
Septic Shock (Infections and infestations) | 0
Sinusitis (Infections and infestations) | 1
Streptococcal infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 11
Viral diarrhoea (Infections and infestations) | 1
Wound infection (Infections and infestations) | 14
Anastomotic leak (Injury, poisoning and procedural complications) | 5
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1
Cement embolism (Injury, poisoning and procedural complications) | 1
Confusion postoperative (Injury, poisoning and procedural complications) | 12
Fall (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1
Incarcerated incisional hernia (Injury, poisoning and procedural complications) | 1
Incision site erythema (Injury, poisoning and procedural complications) | 1
Incision site pain (Injury, poisoning and procedural complications) | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1
Mental status changes postoperative (Injury, poisoning and procedural complications) | 1
Pancreatic leak (Injury, poisoning and procedural complications) | 2
Peripancreatic fluid collection (Injury, poisoning and procedural complications) | 1
Post procedural urine leak (Injury, poisoning and procedural complications) | 1
Postoperative ileus (Injury, poisoning and procedural complications) | 30
Procedural haemorrhage (Injury, poisoning and procedural complications) | 13
Procedural nausea (Injury, poisoning and procedural complications) | 4
Procedural pain (Injury, poisoning and procedural complications) | 4
Procedural vomiting (Injury, poisoning and procedural complications) | 2
Seroma (Injury, poisoning and procedural complications) | 1
Stoma site discomfort (Injury, poisoning and procedural complications) | 1
Stoma site extravasation (Injury, poisoning and procedural complications) | 2
Stoma site ischaemia (Injury, poisoning and procedural complications) | 1
Urostomy complication (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 1
Blood bicarbonate increased (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blood creatinine increased (Investigations) | 2
Blood culture positive (Investigations) | 1
Cholangiogram (Investigations) | 1
Enterococcus test positive (Investigations) | 1
Haematocrit decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 2
Oxygen saturation decreased (Investigations) | 2
Transaminases increased (Investigations) | 0
Troponin increased (Investigations) | 1
Acidosis (Metabolism and nutrition disorders) | 1
Alkalosis (Metabolism and nutrition disorders) | 1
Decreased appetite (Metabolism and nutrition disorders) | 3
Dehydration (Metabolism and nutrition disorders) | 2
Diabetes mellitus (Metabolism and nutrition disorders) | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Electrolyte depletion (Metabolism and nutrition disorders) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypernatraemia (Metabolism and nutrition disorders) | 2
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2
Lactic acidosis (Metabolism and nutrition disorders) | 2
Malnutrition (Metabolism and nutrition disorders) | 4
Metabolic alkalosis (Metabolism and nutrition disorders) | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2
Compartment syndrome (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Akinesia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 2
Chronic inflammatory demyelinating (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Dysarthria (Nervous system disorders) | 1
Encephalopathy (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 2
Intracranial hypotension (Nervous system disorders) | 1
Multiple sclerosis relapse (Nervous system disorders) | 1
Myoclonus (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 1
Sciatica (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Device leakage (Product Issues) | 1
Device occlusion (Product Issues) | 2
Anxiety (Psychiatric disorders) | 0
Depression (Psychiatric disorders) | 1
Hallucination (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 0
Mental status changes (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 43
Bladder spasm (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 2
Oliguria (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 14
Vesical fistula (Renal and urinary disorders) | 1
Ovarian vein thrombosis (Reproductive system and breast disorders) | 1
Penile pain (Reproductive system and breast disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 3
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Skin necrosis (Skin and subcutaneous tissue disorders) | 1
Abdominal cavity drainage (Surgical and medical procedures) | 1
Abscess drainage (Surgical and medical procedures) | 1
Biliary drainage (Surgical and medical procedures) | 1
Nephrostomy (Surgical and medical procedures) | 1
Vascular catheterisation (Surgical and medical procedures) | 1
Wound drainage (Surgical and medical procedures) | 2
Deep vein thrombosis (Vascular disorders) | 6
Distributive shock (Vascular disorders) | 1
Haematoma (Vascular disorders) | 5
Hypertension (Vascular disorders) | 8
Hypotension (Vascular disorders) | 38
Peripheral artery thrombosis (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 2
Shock haemorrhagic (Vascular disorders) | 1
Venous thrombosis (Vascular disorders) | 2
Wound secretion (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03469570/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-25): https://cdn.clinicaltrials.gov/large-docs/70/NCT03469570/SAP_001.pdf